CLINICAL TRIAL: NCT06260657
Title: Search for Olfactory Cells Within the Fetal Ethmoid Epithelium
Acronym: COEF
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, JANKOWSKI Roger, Professor, Central Hospital, Nancy, France
Other Study IDs: 2021PI124
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Fetal Ethmoidal Mucosa
Keywords: Ethmoid; Embryology; Olfaction; Evo-devo; Primary olfactory neurons
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Histological fetal data (analysis focused on the ethmoidal block).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fetal ethmoids
  Interventions: Other: Histological analysis on fetal ethmoids

INTERVENTIONS:
Other: Histological analysis on fetal ethmoids — Immunohistological analysis (immunohistochemical or immunofluorescent) on fetal ethmoids

SUMMARY:
The recent rhinological functional approach known as "Evo-Devo" leads us to consider the nose not as a single organ, but as the construction of a specifically olfactory organ within which functional respiratory structures have developed over the course of species evolution in the same way they develop during human embryogenesis.

In adult humans, the olfactory structures are limited to two narrow regions situated at the upper part of the nasal passages known as olfactory clefts. Nevertheless, phylogenetic evidence indicates that these olfactory clefts are vestiges of an olfactory organ that once occupied the entire ethmoid bone in the front of the skull base.

The hypothesis of this study posits that, during the embryological development of the ethmoid bone, it would initially be covered with olfactory mucosa, which would gradually diminish as the lateral masses of the ethmoid formed, eventually persisting exclusively within the olfactory clefts of the ethmoid by the conclusion of the first trimester (end of organogenesis). Besides their fundamental interest, the results of this study could help understand the still unknown pathogenesis of nasal polyposis, a chronic anosmic disease with a prevalence of 2 to 4% in the French and European population.

This study requires a series of ethmoidal samples from human fetuses at various ages between 7 and 15 weeks of gestational age. Specific immunohistological labeling techniques under standard optical microscopy will be used to search for and quantify olfactory nerve cells within the fetal ethmoidal mucosa.

DETAILED DESCRIPTION:
This research project is based on the hypothesis that olfactory epithelium is present within the mucosa of the lateral ethmoid masses, similar to the olfactory fissures at the beginning of the fetal organogenesis period, gradually disappearing before the end of the first trimester in the lateral ethmoid masses as they form.

This study aims to be descriptive, with the objective of identifying this fetal olfactory epithelium and assessing its distribution changes within the ethmoidal mucosa as fetal age progresses.

The chosen method for conducting this study relies on histological analysis using a standard optical microscope of fetal ethmoids (whole bodies or only the cephalic extremity depending on sample size) to preserve their architecture. Microscopic analysis will be coupled with immunohistochemistry or immunofluorescence techniques to characterize the cells of interest: primary olfactory neurons.

Sample collection will be prospective, with the recruitment of fetuses spread over the course of the study, spanning 18 to 24 months. The anticipated minimum sample size is 20 cases. Intermediate analyses are planned in case of non-contribution of samples or if there are a sufficient number of samples to meet the primary and secondary objectives.

The samples are fetal products obtained from either medical or surgical induced abortion procedures, with a gestational age of a minimum of 7 weeks amenorrhea and up to 14 weeks + 6 days.

Sample recruitment is planned to take place within the Orthogeny Service of the University Hospital Maternity in Nancy, integrated into existing service protocols (medical or surgical abortions), and after clear and fair information and obtaining written informed consent from the patients by the investigators. The relevant healthcare teams are informed of the ongoing research. The impact of the research on patient care should be minimized as much as possible to avoid disrupting the patients' process and the medical procedure being carried out. No treatment protocols should be modified or disturbed by this protocol or, if necessary, by the on-site investigators.

In accordance with the 2021 update of the Good Practice Recommendations provided by the French National Authority for Health (HAS) and validated by the French National College of Gynecology and Obstetrics (CNGOF), every abortion procedure includes a prior medical consultation held within 5 days following a woman's request. This consultation precedes the procedure by a few days and aims to provide information about the procedure itself to the patients and address the clinical and paraclinical medical prerequisites necessary for its successful execution. During this time, there is no intervention by the investigators to respect the proper implementation of the medical procedure, which requires a crucial information period during which interference is preferable to be avoided.

Patient information about the conducted research and obtaining written consent is planned to occur upon the patients' admission to the Outpatient Unit of Gynecology and Obstetrics. This phase, in the form of a brief oral interview following their admission by the medical and paramedical teams, is the responsibility of the investigators. It is documented in a paper document that complies with legal establishment directives, produced in duplicate, with one copy retained by the investigators for the DRCI (Clinical Research and Innovation Department), and the second retained by the patient.

The date of the last menstrual period is recorded by the investigators after the interview. This is the only personal or medical data collected from hospitalized patients. Once the procedure is completed (medical or surgical) according to the medical protocol established by the practitioners in the Orthogeny Service, the expulsion or aspiration products are collected and immediately placed in a sealed biopathological collection container while still fresh.

Each sample is marked with an inclusion number: COEF#N° and the gestational age in weeks calculated from the date of the last menstrual period. These data are systematically indexed in an Excel® spreadsheet on a secure computer in the hospital establishment. The sample is promptly transported by the investigators to the Fetal Pathology Laboratory of the University Hospital Maternity in Nancy for rapid freezing at -80°C. A preliminary examination of the products under a binocular microscope is performed to isolate fetal material of interest: whole bodies, complete or fragmented cephalic extremities, including the intact facial mass.

The conditioning of each sample is planned to be standardized. After the recruitment of 10 cases, frozen samples are subjected to a cryosection procedure using a specific Cryocut® microtome. This step allows the creation of serial sections with a thickness of approximately 5 micrometers, mounted on glass slides. An initial extemporaneous examination phase with standard HES staining enables the precise identification of the ethmoid block and subsequently the creation of a series of coronal sections. At this stage of development, skeletal structures are not ossified, avoiding a decalcification phase. Each produced slide is marked with a "Research Number," computer-assigned and automatically given by the histological analysis software used by the Laboratory: Ariane SX®. These numbers are also indexed electronically in relation to the sample data (COEF#N° and gestational age).

The series of slides thus created are treated with immunohistochemistry or immunofluorescence techniques.

The planned immunohistological markers include: Synaptophysin (SP), Neurospecific Enolase (NSE), Neuronal Cell Adhesion Molecule (NCAM), and Oligodendrocyte Transcription Factor (OLIG2). These markers are known monoclonal antibodies referenced in the literature for identifying mature and immature primary olfactory neurons.

After labeling the slides, they are passed through a photographic scanner to generate a digital file containing all the images obtained for each sample. Each file is titled according to the indexing number of each sample: COEF#N°. The recorded image files bear the corresponding slide " Research " number.

Given the purely descriptive nature of this study, descriptive statistics are planned.

After analysis, each series of slides is physically stored at 4°C in the Fetal Pathology Laboratory under the responsibility of the investigators. At the end of the study, these slides will be grouped for preservation within a dedicated collection at the Lorraine Biological Resources Center.

ELIGIBILITY:
Inclusion Criteria:

* Fetus aged at least 7 weeks of gestation up to 14 weeks + 6 days.
* Fetus resulting from an in-hospital procedure of voluntary termination of pregnancy, either medicinal or surgical.
* Fetus whose mother is of legal age and legally responsible.
* Fetus whose mother has been provided with fair and complete information about the research conducted and has given informed, voluntary, and written consent for the use of fetal products from the voluntary termination of pregnancy procedure she is undergoing.
* Fetus whose mother has not objected to the utilization of data derived from the research.

Exclusion Criteria:

* Fetus macroscopically exhibiting a craniofacial malformation

Ages: 7 Weeks to 15 Weeks | Sex: All
Age Groups: Child
Study Population: Fetus aged 7 to 14+6 weeks of gestational age resulting from an in-hospital voluntary termination of pregnancy procedure
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Immunohistological positive signal of primary olfactive neurons | Once a series of 10 recruited samples is assembled, ca. 10 month

SECONDARY OUTCOMES:
Concentration of primary olfactory neurons immunohistological signals | Once a series of 10 recruited samples is assembled, ca. 10 month
  Concentration within the lateral masses of the ethmoid boneas a function of fetal age

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire - Service ORL, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marquez S, Tessema B, Clement PA, Schaefer SD. Development of the ethmoid sinus and extramural migration: the anatomical basis of this paranasal sinus. Anat Rec (Hoboken). 2008 Nov;291(11):1535-53. doi: 10.1002/ar.20775. PMID 18951481
- [Background] Yee KK, Craven BA, Wysocki CJ, Van Valkenburgh B. Comparative Morphology and Histology of the Nasal Fossa in Four Mammals: Gray Squirrel, Bobcat, Coyote, and White-Tailed Deer. Anat Rec (Hoboken). 2016 Jul;299(7):840-52. doi: 10.1002/ar.23352. Epub 2016 May 2. PMID 27090617
- [Background] Glusman G, Yanai I, Rubin I, Lancet D. The complete human olfactory subgenome. Genome Res. 2001 May;11(5):685-702. doi: 10.1101/gr.171001. PMID 11337468
- [Background] Leopold DA, Hummel T, Schwob JE, Hong SC, Knecht M, Kobal G. Anterior distribution of human olfactory epithelium. Laryngoscope. 2000 Mar;110(3 Pt 1):417-21. doi: 10.1097/00005537-200003000-00016. PMID 10718430
- [Background] Bodino C, Jankowski R, Grignon B, Jimenez-Chobillon A, Braun M. Surgical anatomy of the turbinal wall of the ethmoidal labyrinth. Rhinology. 2004 Jun;42(2):73-80. PMID 15224633
- [Background] Escada PA, Lima C, da Silva JM. The human olfactory mucosa. Eur Arch Otorhinolaryngol. 2009 Nov;266(11):1675-80. doi: 10.1007/s00405-009-1073-x. PMID 19714350
- [Background] Jankowski R, Perrot C, Nguyen DT, Rumeau C. Structure of the lateral mass of the ethmoid by curved stacking of endoturbinal elements. Eur Ann Otorhinolaryngol Head Neck Dis. 2016 Nov;133(5):325-329. doi: 10.1016/j.anorl.2016.07.007. Epub 2016 Aug 5. PMID 27502821
- [Background] Lund VJ, Stammberger H, Fokkens WJ, Beale T, Bernal-Sprekelsen M, Eloy P, Georgalas C, Gerstenberger C, Hellings P, Herman P, Hosemann WG, Jankowski R, Jones N, Jorissen M, Leunig A, Onerci M, Rimmer J, Rombaux P, Simmen D, Tomazic PV, Tschabitscherr M, Welge-Luessen A. European position paper on the anatomical terminology of the internal nose and paranasal sinuses. Rhinol Suppl. 2014 Mar;24:1-34. PMID 24720000
- [Background] Yamagishi M, Nakamura H, Takahashi S, Nakano Y, Iwanaga T. Olfactory receptor cells: immunocytochemistry for nervous system-specific proteins and re-evaluation of their precursor cells. Arch Histol Cytol. 1989;52 Suppl:375-81. doi: 10.1679/aohc.52.suppl_375. PMID 2510793
- [Background] Smutzer G, Lee VM, Trojanowski JQ, Arnold SE. Human olfactory mucosa in schizophrenia. Ann Otol Rhinol Laryngol. 1998 Apr;107(4):349-55. doi: 10.1177/000348949810700415. PMID 9557772
- [Background] Durante MA, Kurtenbach S, Sargi ZB, Harbour JW, Choi R, Kurtenbach S, Goss GM, Matsunami H, Goldstein BJ. Single-cell analysis of olfactory neurogenesis and differentiation in adult humans. Nat Neurosci. 2020 Mar;23(3):323-326. doi: 10.1038/s41593-020-0587-9. Epub 2020 Feb 17. PMID 32066986